CLINICAL TRIAL: NCT05023980
Title: A Phase 3 Open-Label, Randomized Study of Pirtobrutinib (LOXO-305) Versus Bendamustine Plus Rituximab in Untreated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of Pirtobrutinib (LOXO-305) Versus Bendamustine Plus Rituximab (BR) in Untreated Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: BRUIN CLL-313
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18088; J2N-OX-JZNP (Other: Eli Lilly and Company); LOXO-BTK-20023 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: BTKi; BTK Inhibitor; Hematologic Disease; Lymphoma, non-Hodgkin's; Lymphoma, B-cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — pirtobrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 into Arm A and Arm B. Patients randomized to Arm B who have disease progression (PD) confirmed by independent review committee (IRC) may be eligible to crossover into Arm A.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Pirtobrutinib) (Experimental): Pirtobrutinib administered orally
  Interventions: Drug: Pirtobrutinib
- Arm B (BR) (Active Comparator): Bendamustine plus rituximab administered intravenously (IV)
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Pirtobrutinib — Oral
  Other Names: LOXO-305; LY3527727
  Arms: Arm A (Pirtobrutinib)
Drug: Bendamustine — IV
  Other Names: Treanda; Treakisym; Ribomustin; Levact
  Arms: Arm B (BR)
Drug: Rituximab — IV
  Other Names: Rituxan; MabThera; Truxima; Riabni; Ruxience
  Arms: Arm B (BR)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of pirtobrutinib (LOXO-305; Arm A) compared to BR (Arm B) in patients with CLL/SLL who have not been treated. Participation could last up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL requiring therapy, per iwCLL 2018 criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Adequate organ function
* Platelets greater than or equal to (≥)75 x 10⁹/liter (L) (≥50 × 10⁹/L for patients with evidence of bone marrow infiltrate), hemoglobin ≥8 grams/deciliter (g/dL), and absolute neutrophil count ≥0.75 x 10⁹/L
* Kidney function: Estimated creatinine clearance ≥40 milliliters per minute (mL/min)

Exclusion Criteria:

* Known or suspected Richter's transformation at any time preceding enrollment
* Prior systemic therapy for CLL/SLL
* Presence of 17p deletion
* Central nervous system (CNS) involvement
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP])
* Significant cardiovascular disease
* Active hepatitis B or hepatitis C
* Active cytomegalovirus (CMV) infection
* Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection
* Known human immunodeficiency virus (HIV) infection, regardless of cluster of differentiation 4 (CD4) count
* Concurrent use of investigational agent or anticancer therapy except hormonal therapy
* Patients requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist
* Vaccination with a live vaccine within 28 days prior to randomization
* Patients with the following hypersensitivity:

  * Known hypersensitivity, including anaphylaxis, to any component or excipient of pirtobrutinib or bendamustine
  * Prior significant hypersensitivity to rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate progression-free survival (PFS) of pirtobrutinib (Arm A) compared to bendamustine and rituximab (Arm B) | Up to approximately 5 years
  Assessed by blinded independent review committee (IRC) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 Response Criteria

SECONDARY OUTCOMES:
To evaluate the effectiveness of Arm A compared to Arm B: Progression-free survival (PFS) | Up to approximately 5 years
  Assessments of effectiveness include PFS, assessed by investigator
To evaluate the effectiveness of Arm A compared to Arm B: Overall survival (OS) | Up to approximately 5 years
  Assessments of effectiveness include OS, assessed by investigator
To evaluate the effectiveness of Arm A compared to Arm B: Time to next treatment (TTNT) | Up to approximately 5 years
  Assessments of effectiveness include TTNT, assessed by investigator
To evaluate the effectiveness of Arm A compared to Arm B: Overall response rate (ORR) | Up to approximately 5 years
  Assessments of effectiveness include ORR, assessed by investigator and IRC
To evaluate the effectiveness of Arm A compared to Arm B: Duration of Response (DOR) | Up to approximately 5 years
  Assessments of effectiveness include DOR, assessed by investigator and IRC
To evaluate the effectiveness of Arm A compared to Arm B in patient-reported disease-related symptoms | Up to approximately 5 years
  Based on time to worsening of CLL/SLL-related symptoms
To evaluate the effectiveness of Arm A compared to Arm B in patient-reported physical functioning | Up to approximately 5 years
  Based on time to worsening of physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (108):
- United States (5):
  - California Research Institute, Los Angeles, California
  - Innovative Clinical Research Institute, Whittier, California
  - Oncology-Hematology Associates of West Broward, Coral Springs, Florida
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Clinical Research Alliance, Inc., Westbury, New York
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Peninsula Private Hospital, Frankston, Victoria
- Austria (2):
  - Uniklinikum Salzburg, Salzburg
  - Klinik Ottakring, Vienna
- Brazil (5):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado - Mae de Deus Center, Porto Alegre, Rio Grande do Sul
  - Hemocentro Unicamp, Campinas, São Paulo
  - Fundação Doutor Amaral Carvalho, Jaú, São Paulo
- Bulgaria (4):
  - UMHAT "Sveti Georgi" EAD, Plovdiv
  - UMHAT 'Sv. Ivan Rilski', EAD, Sofia
  - "SHATHD" EAD, Sofia, Sofia
  - UMHAT - Prof. Dr. Stoyan Kirkovich" AD, Stara Zagora
- China (19):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyany, Liaoning
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - Shanghai Tongren Hospital, Changning District, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Hangzhou Linping District, Hangzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Henan Cancer Hospital, Zhengzhou
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Hospitalier Le Mans, Le Mans, France
- Hungary (3):
  - Debreceni Egyetem Orvos-es Egészsegtudomanyi Centrum, Debrecen
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Italy (12):
  - Irccs Crob, Rionero in Vulture, Potenza
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda Comitato Etico Milano Area C, Milan
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Azienda Ospedale Maggiore Della Carita, Novara
  - Istituto di Ematologia-C.R.E.O. (Centro di Ricerche Emato-Oncologich), Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - Azienda sanitaria integrata università di Trieste, Trieste
- Japan (11):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Fukui Medical University Hospital, Yoshida-Gun, Fukui
  - Hokuyukai Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Tohoku University Hospital, Sendai, Miyagi
  - NHO Sendai Medical Center, Sendai, Miyagi
  - Dokkyo Medical University - Koshigaya Hospital, Koshigaya, Saitama
  - University of Yamanashi Hospital, Chūō, Yamanshi
  - Aomori Prefectural Centeral Hospital, Aomori
  - JCHO Kyushu Hospital, Fukoka-ken
- New Zealand (4):
  - North Shore Hospital, Haematology Research, Takapuna, Auckland
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Christchurch Hospital, Christchurch
  - Middlemore Clinical Trials, Papatoetoe
- Poland (12):
  - Wojewodzki Szpital Specjalistyczny, Iwaszkiewicza 5, Legnica
  - Klinika Hematoonkologii i Transplantacji Szpiku SPSK1 Lublin, Lublin, Lubelskie V
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Poznan, Skorzewo, Poznan
  - KO-MED Centra Kliniczne, Biała Podlaska
  - Szpital Uniwersytecki nr 1 im. Antoniego Jurasza, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Nasz Lekarz Osrodek Badan Klinicznych, Torun
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Cuire - Państwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny Klinika, Wroclaw
- Portugal (3):
  - Centro Clínico Académico - Braga (2CA-Braga) (Hospital de Braga), Braga
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (4):
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova, Dolj
  - Institutul Clinic Fundeni - Centrul de Hematologie si Transplant Medular, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Institutului Regional de Oncologie IASI, Iași
- Academician I.P. Pavlov First St-Petersburg State Medical University, Saint Petersburg, Russia
- South Korea (6):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - The Catholic University of Korea-Seoul St. Mary's Hospital, Seocho-Gu, Seoul
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Inje Univ Busan Paik Hospital, Busan
- Spain (6):
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid, Comunidad de
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville
- Taiwan (4):
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- Birmingham Heartlands Hospital, Birmingham, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Pirtobrutinib (LOXO-305) Versus Bendamustine Plus Rituximab (BR) in Untreated Patients With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) (BRUIN CLL-313) — https://trials.lilly.com/en-US/trial/302156